CLINICAL TRIAL: NCT01302548
Title: THE EFFECT OF WOUND IRRIGATION WITH IRRISEPT™ Delivery System ON ABSCESS HEALING IN PATIENTS PRESENTING TO THE EMERGENCY DEPARTMENT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not accrue the required number of study subjects.
Sponsor: University of Florida (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20101227
Record Dates: First submitted 2010-09-29; First posted 2011-02-24 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Abscess
Keywords: Abscess; Wound Irrigation; Wound Debridement; Wound Healing; Incision and drainage; Chlorhexidine
MeSH Terms: conditions — Abscess; Surgical Wound | interventions — Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IRRISEPT (Experimental): Device containing sterile water and chlorhexidine gluconate (CHG)
  Interventions: Device: IRRISEPT
- Usual Care (Active Comparator): The usual care method will either be the saline irrigation or incision and drainage depending on the physicians discretion.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Device: IRRISEPT — Device containing sterile water and chlorhexidine gluconate (CHG)
  Arms: IRRISEPT
Procedure: Usual Care — The usual care method will either be the saline irrigation or incision and drainage depending on the physicians discretion.
  Other Names: Saline irrigation; Incision & Drainage
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine if wound cleansing and irrigation using the IRRISEPT Chlorhexidine Gluconate(CHG)solution, applying a given volume with a pressurized stream, will improve the outcome for infected abscesses in patients that present in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent individuals 12 years of age or older with an uncomplicated abscess
* Patient must be able to answer questions and be medically stable as defined by the Emergency Department physician
* Patient must voluntarily participate in the study

Exclusion Criteria:Patients with any of the following are excluded:

* Currently receiving antibiotics or received antibiotics within last 72 hours
* Evidence of systemic infection (fever, aches, chills, nausea)
* Requires admission to the hospital for infection or for any other reason(s)
* Abscess caused by a human or animal bite
* Prior history of hypersensitivity or allergy to Chlorhexidine Gluconate (CHG)
* Immunodeficiency (Examples: HIV Positive, Crohns Disease, Systemic Lupus Erythematosus, Addison's disease, psoriasis, splenectomy, leukemia, cancer on chemotherapy)
* Currently on any immune-modifying medication (Examples: prednisone, antivirals)
* History of chronic skin infection (3 or more in the past year)
* Chronic medical problem, for example end-stage heart, liver, kidney, or lung disease, diabetes mellitus, peripheral vascular disease, history of organ transplant
* Mental illness including but not limited to substance abuse, dementia, schizophrenia or mentally handicapped or challenged
* Incarcerated
* Patient is pregnant or thinks she may be pregnant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Petrik, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IRRISEPT | Usual Care
Started | 14 | 19
Completed | 12 | 18
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IRRISEPT | Usual Care | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.42 (9.04) | 24.83 (9.81) | 27.87 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Abscess Healing Based on Abscess Measurement Scale
Description: The abscess healing process will use two methods: 1) "usual method" includes saline irrigation and/or incision & drainage, and 2) the use of IRRISEPT solution. The Abscess Measurement Scale was measured using a centimeter ruler.
  Scale 8cm - 10cm = Severe 6cm - 8cm = Moderate/severe 4cm - 6cm = Moderate 2cm - 4cm = Mild/moderate 0cm - 2cm = Mild
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IRRISEPT | Usual Care
Number analyzed (Participants) | 12 | 18
units on a scale | 2.750 (0.6216) | 2.833 (0.9852)
Statistical Analysis 1: Comparison: IRRISEPT vs Usual Care; Ho: There is not a significant difference between the use of IRRISEPT solution and the "usual care methods" on abscess healing. This study did not enroll an adequate number of patients to meet sufficient power; Test type: Superiority or Other; p = .7970, t-test, 2 sided — This is unadjusted; Degrees of freedom = 28; Mean Difference (Net) = .0833, 95% CI 2-sided [-.5738 to .7405], Standard Deviation .8609

2. Secondary Outcome: Number of Patients Prescribed Oral Antibiotics
Description: Number of patients prescribed oral antibiotics
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | IRRISEPT | Usual Care
Number analyzed (Participants) | 12 | 18
participants | 1 | 5
Statistical Analysis 1: Comparison: IRRISEPT vs Usual Care; Ho: There is not a significant difference between the proportion of patients requiring antibiotics after the use of IRRISEPT solution vs. the "usual care methods" on abscess healing. This study did not enroll an adequate number of patients to meet sufficient power; Test type: Superiority or Other; p = .3575, Fisher Exact — This is unadjusted; Cell (1,1) Frequency (F) = 13; Odds Ratio (OR) = .2364, 95% CI 2-sided [.0239 to 2.3394]

3. Secondary Outcome: Abscess Measurement Using a Abscess Measurement Scale in Methicillin-resistant Staphylococcus Aureus (MRSA) Positive Patients.
Description: The Abscess Measurement Scale was measured using a centimeter ruler.
  Scale 8cm - 10cm = Severe 6cm - 8cm = Moderate/severe 4cm - 6cm = Moderate 2cm - 4cm = Mild/moderate 0cm - 2cm = Mild
Time Frame: 48 hours
Population: Only participants that were MRSA-positive, were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IRRISEPT | Usual Care
Number analyzed (Participants) | 5 | 1
units on a scale | 2.4 (.5477) | 2.0 (NA) — There was only one patient in this group.
Statistical Analysis 1: Comparison: IRRISEPT vs Usual Care; Ho: There is not a significant difference between the use of IRRISEPT solution and the "usual care methods" on abscess healing in patients that are MRSA positive. This study did not enroll an adequate number of patients to meet sufficient power; Test type: Superiority or Other; p = .5415, t-test, 2 sided — This is unadjusted; Degrees of freedom = 4; Mean Difference (Net) = -.400, 95% CI 2-sided [-2.0659 to 1.2659], Standard Deviation .5477

ADVERSE EVENTS:
Time Frame: 02/26/2011 - 08/09/2012
Arm/Group | IRRISEPT | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 1/14 | 0/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IRRISEPT (N=14) | Usual Care (N=19)
Increased Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Increased pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No